CLINICAL TRIAL: NCT01246817
Title: Evaluation of the Activity of Temsirolimus With FDG-PET and FLT-PET in Patients With Renal Cell Cancer
Brief Title: Temsirolimus-RCC-imaging
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCNONCO200903
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Renal Cell Cancer
Keywords: Carcinoma, Renal Cell; temsirolimus; FLT-PET; FDG-PET; Adult patients with metastatic RCC (any histology and any MSKCC prognostic score), with documented; progressive disease after more than two prior systemic treatments with any of the following: cytokines (±; chemotherapy), sunitinib, sorafenib, or bevacizumab (± IFN).
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Temsirolimus — temsirolimus (standard schedule: 25 mg weekly, by 1-hour i.v. infusion)

SUMMARY:
This study uses one trialdrug: Temsirolimus (sometimes called Torisel ® ). Temsirolimus is an mTOR inhibitor. It is an agent that is specifically aimed at disrupting cell division (needed for cancer cell growth). Temsirolimus has been shown to inhibit the growth of cancer cells. For patients with metastatic kidney cancer Temsirolimus is now a registered , conventional therapy. It has been recorded for patients as they get renal cell cancer metastases and which looks as if the tumor is aggressive.

This is a phase II trial. This means that the investigators look at how effectively temsirolimus is, after treatment with other drugs against kidney cancer. Effective means that the investigators see how well the treatment is, the investigators look at how long the disease is not growing and if it does, that is smaller. The possible side effects will be carefully watched.

DETAILED DESCRIPTION:
The prognosis of metastatic renal cell carcinoma (mRCC) patients has improved the last couple of years, due to the treatment with angiogenesis inhibitors and mTOR inhibitors. First line and second line therapy is nowadays standard. However, responses on third or fourth line therapy, in RCC patients participating in phase I studies have been observed. As yet the optimal sequence of therapeutic agents in mRCC is not known and data on progression free survival of third or fourth line treatment is not available. More and more patients with metastatic RCC will receive multiple sequential treatments. A large proportion of those patients will remain in a good condition and have a good quality of life. Those are the candidates for new lines of therapy.

In the evaluation of new treatments the difficulty lies in the way of assessment of activity of new drugs. In the past, chemotherapy induced real volume responses, whereas with the new targeted agents volume reponse may take a long period of time (more than 6 months is not exceptionial), or will never induce a real decrease in tumor volume, while the patient may benefit from a long period of stable disease. All these new drugs are costly and not without side effects, and therefore there is an urgent need for new end points of therapy, better reflecting the activity of the drug.

In first line poor prognosis metastatic RCC patients mTor inhibition with temsirolimus has become standard therapy based on an improvement in PFS and OS. Also for temsirolimus RECIST criteria have been used. However, by using the RECIST criteria for the evaluation of efficacy only the change in tumour volume is assessed. Temsirolimus is an antiproliferative anti cancer drug and proliferation might be assessed by FLT PET or FDG PET.

Until now only very limited data have been published on the role of FDG PET and FLT PET after mTor inhibitors. FLT PET seems promising in mice glioblastoma in mice treated with mTor inhibitors. Another very recent paper reports the value of FDG PET as suurogate marker of everolimus activity, also in mice. Only one clinical study in which FDG PET was used in patients treated with mTor inhibitors had included patients with a mixture of diagnoses.

Therefore, we propose to investigate in a systematic way whether molecular imaging with FLT-PET and/or FDGPET is a better predictor of response and progression free survival (PFS) than evaluation by standard anatomical imaging by CT-scan in RCC patients treated with temsirolimus. Furthermore, we propose to investigate the optimal way of assessment of molecular characteristics of the tumor (metabolism, proliferation) by comparing FLT-PET with FDG-PET.

ELIGIBILITY:
Inclusion Criteria:

1. patients with histologically confirmed, advanced (stage IV or recurrent disease) RCC who have received at least one prior angiogenesis inhibitor for their disease.
2. Karnofsky performance status ≥ 70.
3. At least 1 measurable lesion that can be accurately measured in at least 1 dimension with the longest diameter ≥ 10-mm when measured by spiral computerized tomography (CT, 5-mm slice thickness contiguous)
4. Age ≥ 18 years.
5. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1500 cells/mm3), platelet count ≥ 100 x 109/ L (100,000 cells/ mm3), hemoglobin ≥ 8.0 g/dL (5.0 mmol/L).
6. Adequate renal function (serum creatinine ≥ 1.5 times the ULN) or creatinin clearance of ≥ 50 ml/min
7. Adequate hepatic function (bilirubin ≤ 1.5 times the ULN, aspartate transaminase (AST) ≤ 3 times the ULN [≤ 5 times the ULN if liver metastases are present]).
8. Fasting serum cholesterol ≤ 350 mg/dL (9.0 mmol/L), triglycerides ≤ 400 mg/dL (4.56 mmol/ L).
9. Subjects receiving cytochrome P450 (CYP) 3A4 inducers or inhibitors must be on stable doses for at least 1 week prior to randomization.
10. Life expectancy of at least 8 weeks.
11. Negative pregnancy test for female patients of childbearing potential
12. Women and men enrolled into this trial must use adequate birth control measures during the course of the trial and must continue for 3 months after the last dose of temsirolimus.
13. Signed and dated written informed consent form

Exclusion Criteria:

1. Subjects with central nervous system (CNS) metastases. Subjects with a prior history of CNS metastases will be eligible if the screening magnetic resonance imaging (MRI)/CT (with contrast) indicates no residual disease.
2. Prior investigational therapy/agents within 2 weeks of randomization.
3. Prior treatment with a mTOR inhibitor
4. History of other prior malignancy in past 5 years, other than basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.
5. Not recovered from prior surgery and/or surgery or radiation therapy within 4 weeks of randomization.
6. Immunocompromised subjects, including subjects known to be human immunodeficiency virus (HIV) positive, hepatitis B positive, or hepatitis C positive.
7. Active infection or serious intercurrent illness.
8. Presence of unstable angina or myocardial infarction within the previous 6 months (prior to screening), use of ongoing maintenance therapy for life-threatening arrhythmia, known pulmonary hypertension, or pneumonitis.
9. Pregnant or nursing women, women who are of childbearing potential who are not using an effective contraceptive method, or men with partners of childbearing potential who are not using an effective contraceptive method. (A woman of childbearing potential is defined as a woman who is biologically capable of becoming pregnant.)
10. Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the FLT-PET and FDG-PET | before and during treatment
  Measurement of 18F-FLT-PET-signal and FDG-PET-signal (ROI analysis and SUVmax calculation), and signal changes during treatment with temsirolimus (percentage change in SUVmax) Correlation of 18F-FLT-PET and FDG-PET before, and signal changes during treatment with treatment outcome (clinical response and PFS).

SECONDARY OUTCOMES:
Progression free survival | after treatment
  Assessment of duration of PFS after treatment with temsirolimus in heavily pre-treated metastatic RCC patients
response rate | during the trial
  Measurement of the response rate
Toxicity | during and after the trial
  patients are monitored during the trial for toxicities using CTC AE version 3.0. If applicable neccesary dose-adjustments will be made
Correlation of pharmacodynamics with PET results | baseline, after 2nd Temsirolimus infusion after the 6th temsirolimus infusion (approx 5 days after), at time of PD and 2 weeks after the last Temsirolimus infusion
  Regulatory T cells, insulin growth factor (IGF), insulin growth factor big protein-2 (IGFBP), angiogenic markers, circulating endothelial cells (CECs) and circulating tumor cells (CTCs) will be determined. The results will be correlated with the PET scanning data.

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, Md PhD, Principal Investigator — University Medical Centre Nijmegen
Locations (1):
- University Medical Centre Nijmegen, Nijmegen, Gelderland, Netherlands